CLINICAL TRIAL: NCT01654614
Title: Diagnostic Capacity of Keratoconus Match Index and Keratoconus Match Probability in Forme Fruste Keratoconus
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Senior Lecturer of Ophthalmology, Democritus University of Thrace
Other Study IDs: 62/18.07.2012
Record Dates: First submitted 2012-07-22; First posted 2012-08-01 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Forme Fruste Keratoconus (FFK)
Keywords: Keratoconus match index; keratoconus probability index; ocular response analyzer; Pentacam; forme fruste keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Forme Fruste Keratoconus Group (FFKG): Forme Fruste Keratoconus Group (FFKG) included patients diagnosed with FFK.
- Control Group (CG): Control group(CG) was formed by refractive surgery candidates.

SUMMARY:
Primary objective of this study was to evaluate the diagnostic capability of keratoconus match index (KMI) and keratoconus match probability (KMP) indexes in forme fruste keratoconus (FFK), and their association with a series of Pentacam-derived keratconus (KC) indexes. KMI and KMP parameters are KC-specifc indexes that are measured by Ocular Response Analyzer (ORA), based on the distinct ORA-derived waveform characteristics of KC eyes.

Study participants were recruited from the Cornea Outpatient service in a consecutive if eligible basis. Two study groups were formed: a) FFK group (FFKG) that included patients diagnosed with FFK, and, b) Control group (CG) was formed by refractive surgery candidates.

All ORA (Reichert Ophthalmic Instrument, Buffalo, NY, USA, software version: 3.01)and Pentacam (Pentacam HR, Oculus Optikgerate GmbH, Heidelberg, Germany)measurements were performed by the same experienced operator in a consistent way

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of keratoconus KC in the fellow eye according to the Amsler-Krumleich criteria (FFKG)
* KISA index between 60 and 100% in the FFK eye (FFKG)
* lack of any KC-related findings / signs in the slit-lamp biomicroscopy (FFKG)
* uneventful ophthalmologic history (CG)
* no indications of corneal pathology in slit-lamp biomicroscopy and Placido disk-based videokeratography (CG)
* KISA index value less than 60% (CG)

Exclusion Criteria:

for both study groups:

* previous incisional eye surgery
* corneal scars and opacities
* history of herpetic keratitis, severe eye dryness
* pregnancy or nursing
* current corneal infection
* glaucoma
* suspicion for glaucoma
* IOP lowering treatment
* underlying autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants were recruited from the Outpatients Cornea service, in a consecutive if eligible basis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Keratoconus Match Index (KMI) | one day
  KMI is the outcome of a neural network calculation of seven ORA-derived waveform scores and represents the similarity of the waveform of the examined eye against the same average waveform scores of the keratoconus eyes in the machine's database.
  Receiver operating characteristics (ROC) curves were applied to determine the overall predictive accuracy of KMI parameter,as described by the area under the curve (AUC), in differentiating FFK cases from normal ones. The impact of Pentacam-derived KC related indexes on KMI was assessed with stepwise forward multivariate regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute of Thrace (ΕΙΤ), Alexandroupoli, Evros, Greece

REFERENCES:
- [Result] Labiris G, Giarmoukakis A, Gatzioufas Z, Sideroudi H, Kozobolis V, Seitz B. Diagnostic capacity of the keratoconus match index and keratoconus match probability in subclinical keratoconus. J Cataract Refract Surg. 2014 Jun;40(6):999-1005. doi: 10.1016/j.jcrs.2013.08.064. Epub 2014 Apr 6. PMID 24713585